# Statistical Analysis Plan

# PRactice of OXYgen Use in COVID-19 patients (PROXY-COVID) – a multicenter observational study

Michela Botta<sup>1</sup>, Oriol Caritg Cirera<sup>2</sup>, David M.P. van Meenen<sup>1</sup>, Anissa M. Tsonas<sup>1</sup>, Willemijn Mooij<sup>1</sup>, Alessia Burgener<sup>1</sup>, Tosca Manriquez<sup>1</sup>, Gentle Sunder Shrestha<sup>3</sup>, Janneke Horn<sup>1,4</sup>, Frederique Paulus<sup>1,5</sup>, Oriol Roca<sup>2</sup>, Marcus J. Schultz<sup>1,6,7,8</sup>

Amsterdam UMC, location University of Amsterdam, Amsterdam, The Netherlands

<sup>1</sup>Department of Intensive Care

Vall d'Hebron University Hospital, Barcelona, Spain <sup>2</sup>Department of Intensive Care

Tribhuvan University of Nepal, Kirtipur, Nepal

3Department of Intensive Care

Amsterdam UMC Research Institute, Amsterdam, The Netherlands

<sup>4</sup>Amsterdam Neuroscience

Amsterdam University of Applied Sciences, Faculty of Health,
Amsterdam, The Netherlands

5ACHIEVE, Centre of Applied Research

Mahidol University, Bangkok, Thailand 
<sup>6</sup>Mahidol–Oxford Tropical Medicine Research Unit (MORU)

University of Oxford, Oxford, United Kingdom

<sup>7</sup>Nuffield Department of Medicine

Hamilton Medical AG, Bonaduz, Switzerland <sup>8</sup>Department of Research and Development

## **Correspondence:**

Michela Botta, MD
Department of Intensive Care
G3–228, Amsterdam UMC, location 'AMC'
Meibergdreef 9, 1105 AZ Amsterdam, The Netherlands
Email: m.botta@amsterdamumc.nl

# **Objectives**

The objective of the study is to compare the amount of supplemental oxygen used with invasive ventilation or noninvasive ventilation (NIV) versus high–flow nasal oxygen (HFNO) in the first 2 days of ventilatory support in patients with acute hypoxemic respiratory failure related to COVID–19.

# **Hypothesis**

The amount of supplemental oxygen used with invasive ventilation or NIV is substantially lower than with HFNO.

## **Patients**

This international study enrolled patients with acute hypoxemic respiratory failure related to COVID-19 that were admitted to the ICUs of two hospitals in the Netherlands and Spain between October 1 2020 and December 31 2020. We excluded patients who received ECMO.

## **Data collected**

- Demographic data and chronic comorbidities were collected at baseline; the Simplified Acute Physiology Score (SAPS) II was calculated using data collected in the first 24 hours after arrival in the ICU. We collected the following data in the first two complete calendar days of ventilation (i.e., ignoring the first calendar day): every 2 hours:
  - o supplemental oxygen mode used, i.e., invasive ventilation, NIV or HFNO
  - o during invasive ventilation and NIV: ventilation mode, inspiratory tidal volume (V<sub>Ti</sub>) (L), total respiratory rate (RR), fraction of inspired oxygen (FiO<sub>2</sub>) (%), positive end-expiratory pressure (PEEP) (cm H<sub>2</sub>O), saturation of

arterial oxygen (SpO<sub>2</sub>) (%), partial pressure of arterial oxygen (PaO<sub>2</sub>) (kPa), and position (supine or prone)

o during HFNO: FiO<sub>2</sub> (%) air flow (L/min), SpO<sub>2</sub> (%), PaO<sub>2</sub> (kPa), and position (supine or prone)

# **Definitions**

Day 1 and Day 2 are the first two complete calendar days of ICU admission and have a duration of 24 hours (from 00:00 to 23:59). Day 0, defined as the time between ICU admission and 23:59 of that day, is ignored.

## **Endpoints**

The primary endpoint is the amount of oxygen used per minute at patient level.

The secondary endpoints are the total amount of oxygen used and the amount of oxygen used per hour at patient level.

The supplemental oxygen per minute (Supplemental Oxygen<sub>min</sub>) is calculated every 2 hours. For invasive ventilation and NIV

Supplemental Oxygen<sub>min</sub> (L) = 
$$V_{Ti}$$
 (L) \* total RR \* (FiO<sub>2</sub> – 0.21)

For the HFNO group

Supplemental Oxygen<sub>min</sub> (L) = air flow (L/min) x (FiO<sub>2</sub> 
$$-$$
 0.21)

Supplemental oxygen per hour (Supplemental Oxygenhour) and total supplemental oxygen on Day 1 and 2 are calculated using the area under the curve (AUC) method.

Statistical analysis plan

Continuous data are reported as medians with interquartile ranges and categorical data as numbers with percentages.

Each patient is assigned to a group named 'invasive ventilation or NIV' and 'HFNO' based on the first used form of ventilatory support, meaning that patients who received HFNO first and invasive ventilation or NIV afterwards is included in the 'HFNO' group and vice versa.

To assess differences between patient groups in both approaches, Wilcoxon-Mann-Whitney test for continuous data and Fisher exact test for categorical data is used. Differences between demographic data, chronic comorbidities and SAPSII are shown in Table 1. Supplemental oxygen per minute (Supplemental Oxygen<sub>min</sub>) at patient level in the two groups is compared using the Wilcoxon-Mann-Whitney. Cumulative frequency distribution of supplemental oxygen per minute are shown for the two groups.

Supplemental oxygen per minute is compared with repeated measures analysis of variance (ANOVA). If significant, a pairwise comparison between every time points is performed.

Sankey diagrams are used to show the different ventilatory support devices used during Day 1 and Day 2.

Supplemental oxygen per hour (Supplemental Oxygenhour) and total supplemental oxygen in the two groups is compared using the Wilcoxon-Mann-Whitney test. Distribution graphs are used to show the differences between the two groups.

In one sensitivity analysis, patients who received both HFNO and invasive ventilation or NIV on Day 1 and Day 2 are excluded, so that patients who received

exclusively HFNO are included in the 'HFNO' group and patients who received only invasive ventilation or NIV are included in the 'invasive ventilation or NIV' group. For this second approach Baseline characteristics are shown in Table 3.

All analyses are conducted in R Studio v. 4.0.3 (R Foundation, Vienna, Austria) and significance level is set at 0.05.